CLINICAL TRIAL: NCT02270541
Title: Single-center Clinical Trial Evaluating the Efficacy, Safety, Feasibility, Reliability, and Cost-effectiveness of In-ambulance Telemedicine for Patients With Suspicion of Acute Stroke
Brief Title: Prehospital Study at the Universitair Ziekenhuis Brussel II
Acronym: PreSSUB II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Research Foundation Flanders (Other); Vrije Universiteit Brussel (Other); Brussels Institute for Research and Innovation (INNOVIRIS) (Unknown); King Baudouin Foundation (Other)
Responsible Party: Principal Investigator, Raf Brouns, MD, PhD, MD PhD, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-003463-38
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Stroke
Keywords: Telemedicine; Prehospital; Emergency Medicine; Stroke
MeSH Terms: conditions — Stroke | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard pre-hospital emergency care by the Paramedic Intervention Team, in accordance with their standing operating procedures.
- Telemedicine (Experimental): In-ambulance teleconsultation by a stroke expert aiming to support the Paramedic Intervention Team by focusing on patient identification, obtaining homeostasis (optimal control of blood pressure, blood oxygenation, temperature, heart rate and rhythm, glycemia), assessment of the patient's neurological status, stroke diagnosis, hospital notification, and patient selection for specific stroke treatment.
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — In-ambulance telemedicine
  Arms: Telemedicine

SUMMARY:
Interventional prospective randomized open blinded end-point (PROBE) single-center clinical trial on the evaluation of the efficacy, safety, feasibility, reliability, and cost-effectiveness of in-ambulance telemedicine for patients with suspicion of acute stroke.

DETAILED DESCRIPTION:
The purpose of PreSSUB II is to evaluate the efficacy, safety, feasibility, reliability and cost-effectiveness of in-ambulance telemedicine during Paramedic Intervention Team transportation of patients with suspicion of acute stroke.

The implementation of expert stroke support in the pre-hospital arena using in-ambulance telemedicine is an innovative approach that opens up new perspectives and allows continuous guidance by a stroke specialist throughout the acute stroke care continuum.

ELIGIBILITY:
Inclusion Criteria:

* Emergency transportation by the Paramedic Intervention Team of the Universitair Ziekenhuis Brussel
* Age >= 18 years
* Suspicion of acute stroke with symptom onset < 12 h or unknown, based on any of the symptoms mentioned in the Belgian manual for medical regulation of pre-hospital care: Hemiparesis, Facial asymmetry, Speech disturbance, Sudden, severe headache, or Confusion.

Exclusion Criteria:

* Patients for whom in-ambulance telemedicine consultation would delay any diagnostic or therapeutic intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Call-to-brain imaging time | within 2 hours
  Interval between emergency call and imaging of the brain by computed tomography or magnetic resonance imaging in the hospital.

SECONDARY OUTCOMES:
Medical events during in-ambulance telemedicine | within 2 hours
  Prevalence of medical events diagnosed and corrected during in-ambulance telemedicine (e.g. blood oxygen desaturation, arterial hypertension, arterial hypotension, hypoglycemia, hyperglycemia, cardiac arrhythmia, decreased level of consciousness, hyperthermia)
Recanalisation therapy | upto 8 hours
  Proportion of patients with ischemic stroke receiving recanalization therapy (i.e. intravenous thrombolysis, endovascular therapy).
Clinical outcome | upto 12 months
  Assessment of the functional status

OTHER OUTCOMES:
Mortality | upto 100 days
  Mortality 90 (± 10) days after stroke
Adverse event | upto 12 months
  In-hospital mortality and any adverse event, in particular known complications of delayed stroke care and thrombolytic therapy (e.g. intracranial hemorrhage, systemic bleeding requiring transfusion, inappropriate use of recanalization therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques De Keyser, MD PhD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Brussels Capital, Belgium